CLINICAL TRIAL: NCT00006231
Title: A Randomized Study to Assess Whether Radiotherapy Prevents Skin Lumps at Sites Where Needles or Tubes Have Been Inserted in Patients With Malignant Mesothelioma
Brief Title: Radiation Therapy in Preventing Metastatic Cancer in Patients Who Have Diagnostic Procedures to Identify Malignant Mesothelioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Glasgow (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068155; CRC-BOC-L52; EU-20033
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2000-10

CONDITIONS: Malignant Mesothelioma; Perioperative/Postoperative Complications
Keywords: localized malignant mesothelioma; advanced malignant mesothelioma; perioperative/postoperative complications
MeSH Terms: conditions — Mesothelioma, Malignant; Postoperative Complications | interventions — Radiotherapy

INTERVENTIONS:
Procedure: quality-of-life assessment
Procedure: standard follow-up care
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known if radiation therapy is effective in preventing metastatic cancer following surgery.

PURPOSE: Randomized phase III trial to determine the effectiveness of radiation therapy in preventing metastatic cancer in patients who have undergone diagnostic procedures to identify malignant mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of radiotherapy in the prevention of metastatic skin nodules or tumor seeding following invasive diagnostic procedures, such as chest drain insertion, pleural aspiration, pleural biopsy, and thoracoscopy, in patients with malignant mesothelioma.
* Determine whether the nodules that develop after radiotherapy are symptomatic in these patients.
* Compare the quality of life of patients treated with radiotherapy vs standard care alone.

OUTLINE: This is a randomized study.

Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive radiotherapy on 3 consecutive days beginning within 3 weeks after chest drain insertion, pleural aspiration, pleural biopsy, or thoracoscopy and once the wounds have healed.
* Arm II: Patients receive standard supportive care alone. Quality of life is assessed at baseline, and then at 1, 2, 4, 6, 9, and 12 months.

Patients are followed at 1, 2, 4, 6, 9, and 12 months.

PROJECTED ACCRUAL: A total of 44 patients (22 per arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven malignant pleural mesothelioma by chest drain insertion, pleural aspiration, pleural biopsy, and/or thoracoscopy within the past 3 weeks

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* At least 3 months

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior systemic chemotherapy for malignant mesothelioma

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior local radiotherapy for malignant mesothelioma

Surgery:

* See Disease Characteristics
* No other invasive procedures to the same chest site during and for 1 year after study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 1998-02; Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Incidence of metastatic skin nodules

CONTACTS AND LOCATIONS:
Overall Officials: Noelle O'Rourke, MD, Study Chair — University of Glasgow
Locations (3):
- United Kingdom (3):
  - West of Scotland Cancer Centre, Glasgow, Scotland
  - Gartnavel General Hospitall, Glasgow, Scotland
  - Stobhill General Hospital, Glasgow, Scotland

REFERENCES:
- [Result] O'Rourke N, Paul J, Hill J: Radiotherapy to mesothelioma drain sites may not be worthwhile: interim report of a randomized study. Lung Cancer 29(1 Suppl 1): A-568, 168, 2000.